CLINICAL TRIAL: NCT03346148
Title: Staff Management About Food Allergy Into ResTaurants in Metz and Strasbourg
Brief Title: Staff Management About Food Allergy Into ResTaurants
Acronym: SMART
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-03Obs-CHRMT
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Food Allergy
Keywords: Food Allergy, Restaurant staff
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of the knowledge levels of restaurant personnel about food allergies. A structured questionnaire was given through a telephonic interview to evaluate the responses of the respondents.

DETAILED DESCRIPTION:
Food allergy is a common disease affecting children and adults in Europe. It's a burden for patients, with an important impact on quality of life. Dining in restaurants may be dangerous for allergic consumers. Currently in France, little training on food allergies is included in the generic food hygiene training that is compulsory for only a minimum of one member of the staff of a restaurant.

ELIGIBILITY:
Inclusion Criteria:

* Etablished in Metz or Strasbourg
* Restaurant staff member

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Restaurant staff member
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
knowledge about food allergy | Day 1
  questionnaire